CLINICAL TRIAL: NCT01313013
Title: A Question Prompt Sheet for Depressive Outpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: PD Dr. Johannes Hamann
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: prompt1
Record Dates: First submitted 2011-03-09; First posted 2011-03-11 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Experimental): question prompt sheet
  Interventions: Behavioral: question prompt sheet
- control (No Intervention): no question prompt sheet

INTERVENTIONS:
Behavioral: question prompt sheet
  Arms: intervention

SUMMARY:
question prompt sheet for outpatients suffering from depression. effects on patient-doctor-communication during the consultation.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* male and female patients
* outpatients
* informed consent

Exclusion Criteria:

* poor German language skills

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)